CLINICAL TRIAL: NCT00343343
Title: A Comparative, Randomised Study With NovoFine® 4 mm Needle Versus NovoFine® 6 mm Needle in Regard to Anatomical Deposition of Sterile Air in Children and Thin Adults With Diabetes and Backflow of Test Medium (Only Adults) After Injection in Thigh and Abdomen
Brief Title: Comparison of NovoFine® Needles (4 mm vs. 6 mm)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PDS322-1749; 2006-000174-78 (EudraCT Number)
Record Dates: First submitted 2006-06-19; First posted 2006-06-22 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 6 mm
Device: NovoFine® needle 4 mm

SUMMARY:
This trial is conducted in Europe. The aim of this investigation is to explore the safety of a 4 mm needle compared to a 6 mm needle when injected in children and lean adults with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Children
* Type 1 diabetes
* Insulin treatment for more than ½ year
* BMI lesser than or equal to 19 kg/m2
* Last HbA1c taken within the last year lesser than 10.5%
* Girls: only prepubertal
* Boys: both pre pubertal and pubertal. Adults
* Type 1 and 2 diabetes
* Insulin treatment for more than ½ year
* BMI lesser than or equal to 23 kg/m2
* Last HbA1c taken within the last year lesser than 10.5%

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products.
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (including country-specific adequate measures, if any).
* Skin disease at abdomen and/or thigh

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Deposition of sterile air depositions.

SECONDARY OUTCOMES:
Thickness of 1) dermis and 2) distance from skin surface to muscle fascia
Amount of backflow

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Denmark (2):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C

REFERENCES:
- [Result] Birkebaek NH, Solvig J, Hansen B, Jorgensen C, Smedegaard J, Christiansen JS. A 4-mm needle reduces the risk of intramuscular injections without increasing backflow to skin surface in lean diabetic children and adults. Diabetes Care. 2008 Sep;31(9):e65. doi: 10.2337/dc08-0977. No abstract available. PMID 18753661
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com